CLINICAL TRIAL: NCT06444854
Title: Patient Reported Outcomes Targeting Early Chest Tube Removal (PROTECTR) Study
Acronym: PROTECTR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Rahul Nayak, Director of Research, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PROTECTR
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Lung Surgery; Chest Tube Removal; Enhanced Recovery After Surgery (ERAS)

STUDY DESIGN:
Intervention Model Description: This study is a single centre, prospective clinical trial evaluating the safety and feasibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Chest Tube Removal (Experimental): early chest tube removal at 3 hours
  Interventions: Procedure: early chest tube removal
- Standard of Care (No Intervention): Routine post operative chest tube care

INTERVENTIONS:
Procedure: early chest tube removal — Chest tube removal
  Arms: Early Chest Tube Removal

SUMMARY:
This study is a single centre, prospective clinical trial evaluating the safety and feasibility of implementing a same day chest tube removal protocol in patients undergoing Video Assisted Thoracic Surgery (VATS) anatomical pulmonary surgery.

DETAILED DESCRIPTION:
Pulmonary resections are performed for a multitude of diagnostic and therapeutic reasons. The last decade has seen a rapid advancement of minimally invasive surgical (MIS) approaches which have resulted in improved patient outcomes. However, the post-operative care pathways have not evolved sufficiently to account for these changes. As such, many patients are still admitted after a minor lung resection for monitoring with a chest tube remaining in situ for a minimum of 24 hours. There have been a few retrospective cohort studies that demonstrate that patients do not experience significant complications during that 24-hour period that would warrant hospitalization. However, there have been no prospective controlled studies evaluating the safety and feasibility of early chest tube removal and discharge after a wedge resection. Furthermore, the maintenance of a large bore chest tube for an extended period is a cause for increased patient discomfort, increased narcotic use and may contribute to chronic pain secondary to intercostal nerve compression. As such, the prolonged chest tube maintenance and hospitalization may overall result in more patient harm than benefit.

Our group recently completed and presented a prospective safety and feasibility study demonstrating that chest tubes can be discontinued as early as 3 hours after minor MIS wedge resections of the lung with no adverse events. This study validated safety criteria that will be implemented moving forward. Furthermore, the maintenance of a large bore chest tube for an extended period is a cause for increased patient discomfort, increased narcotic use and may contribute to chronic pain secondary to intercostal nerve compression. As such, the prolonged chest tube maintenance and hospitalization may overall result in more patient harm than benefit. In the study mentioned previously, early chest tube removal led to 40% more patients being opioid free at post operative day 1 compared to those who underwent routine care.

Nevertheless, it is unclear if patients who undergo more extensive surgeries involving vascular dissection and longer operative times (i.e., pulmonary lobectomies and segmentectomies) will derive the same benefit. The incisions required to complete more complex operations are also larger compared to wedge resections. As such the pain associated with having a chest tube may or may not be as apparent in the setting of the larger incision. It is also unclear what the long-term impact of early chest tube removal has on quality of life in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs or older
* scheduled to undergo elective VATS segmental or lobar resection of the lung

Exclusion Criteria:

* Pulmonary function tests demonstrating forced expiratory volume in 1 second Forced Expiratory Volume (FEV1) <50% predicted, FEV1 <1.5L and/or diffusion lung capacity of carbon monoxide Lung Diffusion Test (DLCO) <50% predicted
* Patient receives an intraoperative pleurodesis
* Conversion to open thoracotomy or mini thoracotomy intraoperatively.
* Underlying cognitive disorder resulting in inability to complete activities of daily living.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of successful same day chest tube removal | 30 days post-op
  These patients have chest tube removed if they meet study criteria
EuroQol 5 Dimension 5 Level (EQ5D5L) score | 30 days post-op
  Difference in EQ5D5L scores between standard care and early chest tube removal on POD1 and POD30.
Mean Morphine Equivalents (MME) Post-Operative Day 1 (POD1) | 24 hours
  Mean Morphine Equivalents used on post operative day 1
Pleural reintervention | 30 days post-op
  Rate of pleural reintervention (defined as requiring reinsertion of a chest tube or return to the operating room)

SECONDARY OUTCOMES:
Complications | 30 days post-op
  The rates of grade 1 to 5 complications as per the Thoracic Surgery Quality Improvement Canada (TSQIC) will be recorded for up to 30 days after surgery in the divisional thoracic REDCap database.
Chest Tube duration | 30 days post-op
  Duration the patient had chest tubes in situ will be measured by collecting the date and time of arrival to Post anesthesia Care Unit (PACU) and the date and time the chest tube was removed.
Unplanned return | 30 days post-op
  Unplanned returns to clinic or emergency room within the first 30 days after surgery
Length Of Stay | 30 days post-op
  Duration of hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Nayak, MD MSc, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No